CLINICAL TRIAL: NCT00374790
Title: Pilot Study to Determine the Efficacy of Iron Supplementation in Preventing the Elevation of Blood Lead Concentrations in Young Children
Brief Title: Iron Supplementation of Lead-exposed Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 0604015
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Lead Toxicity
Keywords: Lead toxicity
MeSH Terms: interventions — ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate

SUMMARY:
The purpose of this study is to compare the efficacy of iron (12.5 mg as ferrous sulfate) and placebo given for 6 months in preventing the elevation of blood lead concentration in children 6-9 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants included if gestational age >36 weeks, birth weight > 2500g, no chronic illness, blood lead concentration <10 mcg/dL, hemoglobin >9 g/dL, zinc protoporphyrin >90 mmol/mol heme
* Mothers included if 18 years or older

Exclusion criteria:

* Hemoglobin >11.5 g/dL

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of blood lead concentrations > 10 mcg/dL
Mean hemoglobin concentration
Mean zinc protoporphyrin concentration

SECONDARY OUTCOMES:
Anthropometry
Oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kordas, PhD, Principal Investigator — Cornell University; Rebecca J Stoltzfus, PhD, Study Chair — Cornell University
Locations (1):
- Clinic for Environmnetal Contaminants, Montevideo, Uruguay